CLINICAL TRIAL: NCT01934114
Title: NIR (Near Infrared Spectral Tomography)Hypoxia Imaging of Breast Tumor Response to Neoadjuvant Chemotherapy in Vivo.
Brief Title: NIR Hypoxia Imaging of Breast Tumor Response to Neoadjuvant Chemotherapy in Vivo
Status: Terminated | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: D1025
Record Dates: First submitted 2013-04-17; First posted 2013-09-04 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2015-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Under Treatment: Patients with locally advanced breast cancer, defined as being clinically appropriate for neoadjuvant therapy
- Normal Cohort: Healthy female volunteers with breast size and epithelial integrity adequate to allow NIR imaging exams

SUMMARY:
The purpose of this study is to determine whether an experimental alternative imaging method, Near Infrared Spectroscopy (abbreviated as NIR), can be used with a controlled respiratory system to examine the breasts for cancer. The NIR system uses light beams to produce an image or picture of the inside of the breast. The respiratory system will help researchers get more information about the breast tissue by changing the amount of oxygen the tissue receives during NIR imaging.

ELIGIBILITY:
Inclusion Criteria:

* NORMAL cohort

  1. Breast size and epithelial integrity adequate to allow NIR imaging exams
  2. No serious associated psychiatric illnesses
  3. Female, ≥25 and <76 years old
  4. Written informed consent
* UNDER TREATMENT cohort

  1. Locally advanced breast cancer, with or without metastatic disease, defined as being clinically appropriate for neoadjuvant therapy
  2. Breast size and epithelial integrity adequate to allow NIR imaging exams
  3. No serious associated psychiatric illnesses
  4. Female, ≥25 and <76 years old
  5. Written informed consent

Exclusion Criteria:

* both cohorts

  1. Pre-existing respiratory conditions:

     1. severe chronic obstructive pulmonary disease (including chronic bronchitis and/or emphysema)
     2. Other respiratory or lung conditions which would place the patient at risk
     3. presence of any other significant cardiac or pulmonary symptoms, such as moderate or severe dyspnea on exertion, orthopnea, or paroxysmal nocturnal dyspnea
  2. Congestive heart failure
  3. Intolerance of hyperoxia or hypercarbia as delivered by the RespirAct breathing circuit
  4. Pregnancy

Ages: 25 Years to 76 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Females with locally advanced breast cancer defined as being clinically appropriate for neoadjuvant therapy and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2010-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Quantify tumor oxygenation response in patients imaged.Determine capability of imaging dynamic to capture oxygenation changes within the tumor. | 18 weeks approximately
  Analyze captured data from use of dynamic NIR topographic oximetry (in a cohort of women receiving conventional anthracycline/taxane based adjuvant chemotherapy).Quantify pathological and clinical outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States